CLINICAL TRIAL: NCT01663493
Title: Randomized Trial Comparing 2 Needles During EUS-FNA of Solid Pancreatic Masses
Brief Title: Comparing Methods to Biopsy Pancreas Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Linda S. Lee, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-P-000955/1
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pancreas Mass Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fine needle aspiration needle (Other): standard Beacon FNA needle
  Interventions: Procedure: FNB
- fine needle biopsy needle (Other): SharkCore fine needle biopsy needle
  Interventions: Procedure: FNB

INTERVENTIONS:
Procedure: FNB

SUMMARY:
This study will examine whether there is any difference in number of passes needed to diagnose pancreatic masses during endoscopic ultrasound-guided biopsies using 2 different types of needles.

ELIGIBILITY:
Inclusion Criteria:

* adult
* pancreas mass

Exclusion Criteria:

* coagulopathy
* mass not approachable by endoscopic ultrasound biopsy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
number of passes | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Linda S Lee, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States